CLINICAL TRIAL: NCT03800212
Title: Study of Survival and Description of Care for Patients With Degenerate Vaterian Ampulloma
Brief Title: Survival and Description of Care for Patients With Degenerate Vaterian Ampulloma
Acronym: AMPULLOMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Other Study IDs: AMPULLOMA COHORT
Record Dates: First submitted 2018-12-31; First posted 2019-01-11 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Ampullary Adenocarcinoma
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: treatment for ampullary adenocarcinoma — all patients treated for ampullary adenocarcinoma (particularly survival without recurrence and prognostic indicators for excised tumours and the duration of disease control for tumours treated with palliative chemotherapy).
  Other Names: no other intervention name to add

SUMMARY:
A Vater's ampulloma is a rare digestive tumour which accounts for under 1% of all digestive tumours. The only curative treatment is complete excision (surgical or endoscopic) of the lesions which is possible in 80% of cases , with or without adjuvant treatment. The reference radical treatment is cephalic duodenopancreatectomy (CDP). The indication for adjuvant treatment is still debated: in view of the aggressive nature of the disease and the high recurrence rate, it would appear appropriate to offer adjuvant treatment, although several studies have failed to find any benefit on survival with post-operative radio-chemotherapy, the most widely studied treatment at present, compared to excision alone. At present there are no phase II studies specifically examining medical treatment of degenerated, inoperable Vater's ampullomas. Some groups propose chemotherapies with 5-FU or gemcitabine, analogous to the treatments used for intestinal, pancreatic or biliary tumours, although neither one has been shown to date to be superior to the other, nor have decision-making criteria been clearly established.In conclusion, a national cohort study is proposed to undertake a prospective analysis of the outcome of all patients treated for ampullary adenocarcinoma (particularly survival without recurrence and prognostic indicators for excised tumours and the duration of disease control for tumours treated with palliative chemotherapy). The treatment methods will be left to the free choice of the investigator and all patients may be included, regardless of stage of their disease. In this study, freezing of tumour fragments is encouraged, as this cohort will be supplemented by a later biological study. In order to recruit sufficient patient numbers, the study will be based on participation of the cooperative groups involved in the management of digestive cancers.

DETAILED DESCRIPTION:
A Vater's ampulloma is a rare digestive tumour which accounts for under 1% of all digestive tumours. In terms of incidence, it is the 3rd most common biliary tract tumour after gallbladder cancer and common bile duct cancer. The incidence of ampullary adenocarcinoma is not well known although it is estimated to be around 0.49 per 100,000 people. The known risk factors are familial adenomatous polyposis (FAP) and Gardner's syndrome, HNPCC (Hereditary Non-Polyposis Colorectal Cancer) syndrome, Peutz-Jeghers syndrome, Crohn's disease and coeliac disease.

Except in its highly localised forms, ampulla of Vater carcinoma carries a poor prognosis. It is a highly lymphophilic disease which commonly metastasises, particularly to the lymph nodes and liver. The prognosis is however considerably better than that of pancreatic adenocarcinoma. In one study which compared 71 ampullomas with 144 adenocarcinomas of pancreatic head, the 5-year survival was 60% for the ampullary carcinomas compared to 20% for pancreatic adenocarcinomas.

More generally, the 5-year survival rate in the literature is between 40-60% and, depending on the study, 10-year survival is approximately 38% .

The only curative treatment is complete excision (surgical or endoscopic) of the lesions which is possible in 80% of cases , with or without adjuvant treatment. The reference radical treatment is cephalic duodenopancreatectomy (CDP). The 5-year survival rate in cases of adenocarcinoma excised by CPD is in the region of 50%, rising to 60-70% if no lymph node invasion is present, compared to 30% when lymph nodes are invaded and median survival is approximately 4.5 years .

The indication for adjuvant treatment is still debated: in view of the aggressive nature of the disease and the high recurrence rate, it would appear appropriate to offer adjuvant treatment, although several studies have failed to find any benefit on survival with post-operative radio-chemotherapy, the most widely studied treatment at present, compared to excision alone . There is only one single randomised study comparing these two forms of management, which shows no benefit in terms of 2 and 5-year survival, although only a small number of patients had an ampullary tumour in this study . The conclusions of several retrospective studies are more subtle, showing results in favour of adjuvant treatment in patients with lymph node disease or a large tumour (T3/T4) .

Some groups have tested the merits of peroperative irradiation. It would appear that this technique does not improve survival, although data on this subject are extremely patchy .

Administration of exclusive adjuvant chemotherapy has been examined in a single randomised study. In this phase III study (ESPAC 3), median overall survival of patients who received adjuvant chemotherapy with FUFOL Mayo for 6 months (n=101) or gemcitabine (n=98) was not significantly improved compared to survival in patients undergoing surgery and not receiving complementary treatment (57.1 versus 43 months, HR= 0.85, p=0.32). A subgroup analysis suggested that the benefit of chemotherapy could be greater in the subgroup of patients with RO resection (p= 0.057, 91% of cases).

Mean survival in patients suffering inoperable tumours is between 9 and 20.4 months depending on the study .

It should be noted however that most of these studies have included tumours other than ampullomas (particularly small bowel adenocarcinomas), making it more difficult to interpret these results, and also that many are old results dating from before the era of modern chemotherapies.

At present there are no phase II studies specifically examining medical treatment of degenerated, inoperable Vater's ampullomas. Some groups propose chemotherapies with 5-FU or gemcitabine, analogous to the treatments used for intestinal, pancreatic or biliary tumours, although neither one has been shown to date to be superior to the other, nor have decision-making criteria been clearly established. One phase II study published in 2009 proposed CAPOX as the reference treatment in light of the promising results obtained. Patients suffering from ampullary cancer in this study however were combined with patients who were suffering from small bowel adenocarcinoma.

In conclusion, a national cohort study is proposed to undertake a prospective analysis of the outcome of all patients treated for ampullary adenocarcinoma (particularly survival without recurrence and prognostic indicators for excised tumours and the duration of disease control for tumours treated with palliative chemotherapy). The treatment methods will be left to the free choice of the investigator and all patients may be included, regardless of stage of their disease. In this study, freezing of tumour fragments is encouraged, as this cohort will be supplemented by a later biological study. In order to recruit sufficient patient numbers, the study will be based on participation of the cooperative groups involved in the management of digestive cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Histologically-proven adenocarcinoma of the ampulla of Vater which is operable or with locoregional or metastatic recurrence after excision less than 6 months previously.

Exclusion Criteria:

* Patients who cannot be followed up regularly for psychological, social, family or geographical reasons.
* Non-ampullary tumours.
* Non-adenocarcinomatous ampullary tumours.
* Ampullary adenocarcinomas which are metastatic or locally advanced from the outset and inoperable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients treated for ampullary adenocarcinoma (particularly survival without recurrence and prognostic indicators for excised tumours and the duration of disease control for tumours treated with palliative chemotherapy).
Sampling Method: Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The time interval between the date of diagnosis of the disease and date of death (all causes). Patients who are alive will be censured at the date of last news.

SECONDARY OUTCOMES:
RECURRENCE FREE SURVIVAL | 3 years
  The time interval between the date of diagnosis of the disease and the date of the recurrence or death (all causes). Patients who are alive without recurrence will be censured at the date of last news.
PROGRESSION FREE SURVIVAL | 5 years
  Time interval between the date of starting treatment and the date of first progression (local or remote, clinical or radiological) or death (all causes). Patients who are alive without progression will be censured at the date of last news. Radiological progression will be defined according to RECIST version 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Julien TAIEB, Principal Investigator — Federation Francophone de Cancerologie Digestive
Locations (36):
- France (36):
  - Ch D'Abbeville, Abbeville
  - Chu Hotel Dieu, Angers
  - Ch Annecy Genevois, Annecy
  - Ch Cote Basque, Bayonne
  - Clinique Champeau, Béziers
  - Chu Saint Andre, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Chu Estaing, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Ch - Sud Francilien, Corbeil-Essonnes
  - Chu Francois Mitterrand, Dijon
  - Chd Vendee, La Roche-sur-Yon
  - Le Kremlin Bicetre, Le Kremlin-Bicêtre
  - Chu Claude Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Ch Nord Essonne, Longjumeau
  - Chu La Croix Rousse, Lyon
  - Hcl Edouard Herriot, Lyon
  - Hcl Pierre Benite, Lyon
  - Hopital de La Timone, Marseille
  - Hopital Saint Joseph, Marseille
  - CH MACON, Mâcon
  - Ch de Meaux, Meaux
  - Chu Caremeau, Nîmes
  - Chr Orleans, Orléans
  - Chu Avicenne, Paris
  - Chu Cochin, Paris
  - Chu La Pitie Salpetriere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Ch Saint Jean, Perpignan
  - CHU Hôpital de la Milétrie, Poitiers
  - Ch Cornouaille, Quimper
  - CH, Reims
  - Ch Saint Malo, St-Malo
  - CLINIQUE, Strasbourg
  - Ch Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: FFCD page — http://www.ffcd.fr/index.php/essais-therapeutiques/pancreas/283-ampullome